CLINICAL TRIAL: NCT05886764
Title: Randomized Trial of Recruitment Strategies for Early Phase Therapeutic Cancer Trials
Brief Title: Novel Outreach Methods to Increase Enrollment to Early Phase Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB23-0221
Record Dates: First submitted 2023-03-03; First posted 2023-06-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Malignancy; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Community-Institutional Relations

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient participants will not be informed of which intervention they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (No Intervention) (No Intervention): Patient participants in this arm will receive no intervention but will be approached by their providers for participation in treatment clinical trials as per the usual methods.
  Provider participants will receive information on available clinical trials for which their patient participant may be eligible from study staff per usual methods. Provider participants will be asked to complete surveys.
- Arm 2 (Digital Intervention) (Experimental): Patient participants in this arm will receive digital messages (email, text, etc.) which include general educational information about clinical trials and available resources.
  Provider participants will also receive digital messages with educational materials and will receive information on available clinical trials for which their patient participant may be eligible from study staff per usual methods. Provider participants will be asked to complete surveys.
  Interventions: Other: Digital Intervention
- Arm 3 (Digital Intervention + Community Outreach) (Experimental): Patient participants in this arm will receive digital messages (email, text, etc.) which include general educational information about clinical trials and available resources. They will also be invited to contact a Community Ambassador for further information and support in the decision to participate in a clinical trial.
  Provider participants will also receive digital messages with educational materials and will receive information on available clinical trials for which their patient participant may be eligible from study staff per usual methods. Provider participants will be asked to complete surveys.
  Interventions: Other: Digital Intervention; Other: Community Outreach

INTERVENTIONS:
Other: Digital Intervention — Digital messages (email, text, etc.) which include general educational information about clinical trials and available resources.
  Arms: Arm 2 (Digital Intervention); Arm 3 (Digital Intervention + Community Outreach)
Other: Community Outreach — Invitation to contact a Community Ambassador for further information and support in the decision to participate in a clinical trial.
  Arms: Arm 3 (Digital Intervention + Community Outreach)

SUMMARY:
This trial will study different outreach methods to assess impact on enrollment of underrepresented minorities (specifically African Americans) to early phase cancer clinical treatment trials. Both patients and providers (those seeing enrolled patients) will be enrolled and receive the study interventions or no intervention (control arm).

ELIGIBILITY:
Inclusion Criteria for Patient Subjects:

* Aged 18 years or older
* Self-described African American race (patients who self-describe as "more than one race" will be included)
* Scheduled for new or consult oncology appointment at the study site
* Scheduled for return outpatient oncology appointment at the study site with a biopsy or radiology encounter within 2 weeks prior to provider visit.

  * for prostate cancer patients: 2 or more increasing prostate specific antigen (PSA) values i the 6 months prior to visit
* other patient identified by research team as potentially having a change in treatment prior to next outpatient oncology appointment at the study site

Inclusion Criteria for Provider Subjects:

* oncology provider at study site scheduled to see patients meeting criteria above

Exclusion Criteria for Patient Subjects:

* Estimated glomerular filtration rate (GFR) less than 30 ml/min/1.73m2 documented within last 2 months and without documented resolutions
* Bilirubin greater than 3.0 ng/dl documented within last 2 months and without documented resolution
* Initiated new anti-cancer therapy within last 2 months
* Evaluated for possible enrollment/randomization in the last 2 months
* Prior enrollment/randomization on this recruitment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that enroll to early phase cancer treatment clinical trials. | within 2 months of randomization

SECONDARY OUTCOMES:
Number of successfully completed outreach efforts | after 30 participants are enrolled to each of arms 2 and 3
Percentage of patients that enroll to early phase cancer treatment clinical trials post intervention. | 2 years from randomization
Percent change in number of African Americans that enroll to cancer clinical trials | 2 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States